CLINICAL TRIAL: NCT01653132
Title: Randomized Double Blind Placebo Controlled Cross-Over Study of Incobotulinum Toxin A (Xeomin®) for Troublesome Sialorrhea in Parkinson's Disease (PD)/Parkinsonism
Brief Title: Incobotulinum Toxin A (Xeomin®) for Troublesome Sialorrhea in Parkinson's Disease (PD)/Parkinsonism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Pushpa Narayanaswami, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2011P00304
Record Dates: First submitted 2012-07-25; First posted 2012-07-30 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Sialorrhea
Keywords: PD
MeSH Terms: conditions — Sialorrhea | interventions — incobotulinumtoxinA; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Incobotulinum Toxin A (Experimental): Twenty units (0.2 ml) of incobotulinum toxin A injected into each parotid gland and 30 units (0.3 ml) to each submandibular gland for a total dose of 100 units using anatomical landmarks
  Interventions: Drug: Incobotulinum Toxin A
- Placebo (Placebo Comparator): Sterile, preservative free 0.9% saline, 1 ml, was used as placebo, and injected into the parotid (0.2 ml each) and submandibular (0.3ml each) glands .
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Incobotulinum Toxin A — Twenty units (0.2 ml) of incobotulinum toxin A were injected into each parotid gland and 30 units (0.3 ml) to each submandibular gland for a total dose of 100 units using anatomical landmarks
  Other Names: Xeomin
  Arms: Incobotulinum Toxin A
Drug: Placebo — Sterile, preservative free 0.9% saline, 1 ml, was used as placebo, and injected into the parotid (0.2 ml each) and submandibular (0.3ml each) glands .
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This study is being conducted this study to determine whether injections of Xeomin®, a type of botulinum toxin into the glands that produce saliva (one pair just below and in front of the ear and the other just under the jaw line) are safe and effective to treat excessive saliva, or drooling in patients with Parkinson's Disease (PD)/parkinsonism.

DETAILED DESCRIPTION:
Participants will be recruited if they have Parkinson's disease, Parkinsonism. Inclusion and exclusion criteria are summarized below. Participants will be screened at the first visit to make sure they are eligible for the trial. They will then undergo baseline testing including neurologic evaluation, questions to assess their memory and cognitive status and evaluation of their disease status using parts of the Unified Parkinsons's Disease Ratings Scale (UPDRS) that are routinely used to follow disease progression. They will be given a questionnaire to evaluate the severity of their drooling. Their saliva production will be measured by having them spit into a cup for 5 minutes, twice.

At the first visit, after making sure they are eligible for the study and performing the baseline testing and procedures, they will be given either Xeomin or placebo (saline injections without medication) injections in the 4 glands that produce saliva. They will not know which injection they received. This visit will take about 2 hours. They will be followed up every month and asked about side effects, have neurologic evaluation and UPDRS testing and fill-in the questionnaire for drooling severity. Saliva volume will be measured as done at the first visit. At either Month 4 or 5, participants will receive the second injection. This will be a "cross-over" injection, i.e., if they received Xeomin at the first injection they will receive saline at the second and vice versa. Thus, all participants will receive the study medication Xeomin, either as the first injection or the second injection at 4 months or 5 months. The follow up after the second injection will be one monthly visit for 3 months, with similar evaluations as described above. The follow-up visit will take about 1 hour each.

ELIGIBILITY:
Inclusion Criteria:

* For PD/ Parkinsonism: 1. PD, Multiple Systems Atrophy (MSA), or Progressive Supranuclear Palsy (PSP) diagnosed by clinical criteria, ages 20-80 with troublesome sialorrhea as defined below**.

  * Sialorrhea that patients or their families or treating physicians think is troublesome

    1. Swallowing function: Functional Oral Intake Scale (FOIS)* of 5 or greater
    2. If patients have been treated with other medications for sialorrhea earlier, they should be off the medications at least 4 weeks prior to the baseline evaluation.
    3. If they are on other medications for sialorrhea at the time of the baseline evaluation, the doses will be held stable throughout the period of the study.
    4. Women of child bearing age will need to be on a reliable method of birth control for the duration of the study.

Exclusion Criteria:

* For PD:

  1. Current use of Coumadin
  2. Concurrent significant medical illness
  3. History of myasthenia gravis or Lambert-Eaton Syndrome
  4. Ongoing substance abuse
  5. History of unreliable follow-up
  6. Past use of Xeomin® or other botulinum toxin preparations
  7. Cognitive impairment, defined as a score ≤ 23/30 on the Mini Mental Status Exam

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pushpa Narayanaswami, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with Parkinson's disease/ parkinsonism with troublesome sialorrhea were recruited from the Movement Disorders clinic at Beth Israel Deaconess Medical Center, Boston, and by providing information to neurologists around the Boston area. Ten subjects were recruited between 9/5/2012 and 2/26/2014. The last study visit was completed on 9/5/14
Pre-assignment Details: 17 subjects were assessed; 7 were excluded because they did not meet study criteria. This was a cross over study; all subjects received both placebo and Incobotulinum toxin injections and were followed up for 3 months after each injection. Washout period was 1-2 months, saliva weight had to be ≥ (baseline- 0.5 SD), to receive the second injection
Groups:
- Placebo First, Then Incobotulinum Toxin A: sterile, preservative free 0.9% saline, 1 ml of saline into the parotid and submandibular glands in first intervention period
- Incobotulinum Toxin A First, Then Placebo: Incobotulinum toxin, 100 units, diluted in 1 ml 0.9% sterile saline. 20 units (0.2 ml) were injected into each parotid gland and 30 units (0.3 ml) into each submandibular gland using anatomical landmarks
Period: First Intervention
Arm/Group | Placebo First, Then Incobotulinum Toxin A | Incobotulinum Toxin A First, Then Placebo
Started | 5 | 5
Completed | 4 (one dropped out: wanted to start anticholinergic drug for tremor that could affect saliva volume) | 5
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Washout 1-2 Months
Arm/Group | Placebo First, Then Incobotulinum Toxin A | Incobotulinum Toxin A First, Then Placebo
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo First, Then Incobotulinum Toxin A | Incobotulinum Toxin A First, Then Placebo
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Ten subjects were recruited; nine completed both periods of the study. One subject dropped out after the first injection because he wanted to start anticholinergics for symptomatic treatment of tremor, and this was an exclusion criterion. His data was excluded.
Groups:
- All Study Participants: Participants who received either Placebo, 1ml of preservative free sterile 0.9% saline, injected into the parotid (0.2 ml each) and submandibular ( 0.3 ml each), or Incobotulinum Toxin A 100 units, 20 units (0.2 ml) of Inco-A were injected into each parotid gland and 30 units (0.3 ml) to each submandibular gland using anatomical landmarks
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9
UPDRS [Median (Inter-Quartile Range); unit: units on a scale] — Unified Parkinsons Disease Rating Scale. The UPDRS is a rating tool to follow the longitudinal course of Parkinson's Disease. It is made up of the 1) Mentation, Behavior, and Mood, 2) Activities of Daily Living and 3) Motor sections. These are evaluated by interview. We used UPDRS, Part 2 Questions 5,6,7 evaluating speech, salivation and swallowing and Part 3 questions 18 and 19 for motor examination of speech and facial expression. The scores for these sections were summed to obtain the total score. The range possible is 0- 20, with 20 reflecting worse disability
  units on a scale | 8.4 [7 to 9]
DFSS [Median (Inter-Quartile Range); unit: units on a scale] — Drooling Frequency and Severity Score:
  The Drooling Score equals the sum of the Severity and Frequency sub-scores.The total score ranges from 2 to 9, with higher scores indicating more severe and frequent drooling
  Drooling Severity Scale
  1. = Never drools, dry
  2. = Mild-drooling, only lips wet
  3. = Moderate- drool reaches the lips and chin
  4. = Severe- drool drips off chin & onto clothing
  5. = Profuse- drooling off the body and onto objects (furniture, books)
  Drooling Frequency Scale
  1. = No drooling
  2. = Occasionally drools
  3. = Frequently drools
  4. = Constant drooling
  units on a scale | 6 [6 to 7]
saliva weight [Mean (Standard Deviation); unit: gms] | 2.13 (4.19)

OUTCOME MEASURES:

1. Primary Outcome: Objectively Measured Salivary Weight
Description: Change in saliva weight between baseline and one month post-injection in the Incobotulinum toxin A period compared to the placebo period.
Time Frame: baseline and one month post-injection in the Incobotulinum toxin A period compared to the placebo period
Measure: Mean (Standard Deviation); unit: gm
Groups:
- Placebo: Sterile, preservative free 0.9% saline, 1 ml, injected into the parotid (0.2 ml each) and submandibular (0.3ml each) glands .
- Incobotulinum Toxin A: Inco-A, 100 units was reconstituted with 1 ml 0.9% sterile saline (dilution: 10 units/0.1 ml). Twenty units (0.2 ml) of Inco-A were injected into each parotid gland and 30 units (0.3 ml) to each submandibular gland using anatomical landmarks
Arm/Group | Placebo | Incobotulinum Toxin A
Number analyzed (Participants) | 9 | 9
gm | -0.07 (1.21) | -0.68 (2.4)
Statistical Analysis 1: Comparison: Placebo vs Incobotulinum Toxin A; Based on the primary outcome measure of mean reduction in saliva weight at 1 month post Inco-A /placebo as compared to baseline, using paired t-test with a two-sided nominal significance (alpha) of 0.05, assuming a correlation of 0.5 between observations, a sample size of 10 pairs has a power of 0.803 to detect a 50% difference in salivary weight; Test type: Superiority or Other; Mean Difference (Net) = -0.194, 95% CI 2-sided [-0.71 to 0.32], Standard Deviation 0.61 — negative values correspond to a reduction in saliva weight with Inco-A

2. Primary Outcome: Objectively Measured Percentage Salivary Weight
Description: Percentage change in saliva weight between baseline and one month post-injection in the Incobotulinum toxin A period compared to the placebo period.
Time Frame: baseline and one month post-injection in the Incobotulinum toxin A period compared to the placebo period
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo | Incobotulinum Toxin A
Number analyzed (Participants) | 9 | 9
percentage change from baseline | -7 (121) | -67 (239)
Statistical Analysis 1: Comparison: Placebo vs Incobotulinum Toxin A; Test type: Superiority or Other; Mean Difference (Net) = -22.3, 95% CI 2-sided [-50.8 to 6.2], Standard Deviation 0.34 — negative numbers represent reduction in saliva weight with Inco-A

3. Secondary Outcome: Change in Drooling Frequency and Severity Scale (DFSS) Scores
Description: measured between baseline and one month post-injection in the Incobotulinum toxin A period compared to the placebo period.Drooling Frequency and Severity Score. The Drooling Score equals the sum of the Severity and Frequency sub-scores. The range is 2-9, higher numbers represent worse drooling Drooling Severity Scale
  1. = Never drools, dry
  2. = Mild-drooling, only lips wet
  3. = Moderate- drool reaches the lips and chin
  4. = Severe- drool drips off chin & onto clothing
  5. = Profuse- drooling off the body and onto objects (furniture, books) Drooling Frequency Scale
  1. = No drooling 2. = Occasionally drools 3. = Frequently drools 4. = Constant drooling
Time Frame: baseline and one month post-injection in the Incobotulinum toxin A period compared to the placebo period
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Incobotulinum Toxin: Incobotulinum Toxin 100 units diluted in 1 ml of sterile 0.9% saline injected in the parotid (20 units, 0.2 ml each)and submandibular (30 units, 0.3ml each) glands of subjects
- Placebo: Placebo: 1ml of preservative free sterile 0.9% saline, injected into the parotid (0.2 ml each)and submandibular ( 0.3ml each) glands of subjects
Arm/Group | Incobotulinum Toxin | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale | -1 (1.41) | -0.67 (0.7)
Statistical Analysis 1: Comparison: Incobotulinum Toxin vs Placebo; Test type: Superiority or Other; Median Difference (Net) = -0.33, 95% CI 2-sided [-1.16 to 0.69], Standard Deviation 1.41 — negative values represent reduction in scores (improvement in drooling) with Inco-A

4. Secondary Outcome: Number of Participants With Response, Defined as Subjects With ≥ 2 Point Improvement in the DFSS Scores.
Description: measured between baseline and one month post-injection in the Incobotulinum toxin A period compared to the placebo period.
Time Frame: baseline and one month post-injection in the Incobotulinum toxin A period compared to the placebo period
Measure: Number; unit: participants
Arm/Group | Incobotulinum Toxin A | Placebo
Number analyzed (Participants) | 9 | 9
participants | 2 | 1
Statistical Analysis 1: Comparison: Incobotulinum Toxin A vs Placebo; Test type: Superiority or Other; Risk Difference (RD) = -0.333, 95% CI 2-sided [-0.633 to 0.071]

5. Secondary Outcome: Number of Participants With Response, Defined as Subjects With ≥ 20% Reduction in Saliva Volume.
Description: as for outcome 4
Time Frame: between baseline and one month post-injection in the Incobotulinum toxin A period compared to the placebo period
Measure: Number; unit: participants
Arm/Group | Incobotulinum Toxin | Placebo
Number analyzed (Participants) | 9 | 9
participants | 3 | 2
Statistical Analysis 1: Comparison: Incobotulinum Toxin vs Placebo; Test type: Superiority or Other; Risk Difference (RD) = -0.11, 95% CI 2-sided [-0.46 to 0.28]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for each subject at monthly visits for the duration of the study, 7-8 months per subject
Description: all subjects were asked at each monthly visit if they had experienced any adverse events since the previous visit. If they responded yes, a checklist of common and rare side effects was used to query subjects, their adverse events were recorded in a standardized fashion and reported to the Committee for Clinical Investigations as per regulations
Groups:
- Incobotulinum Toxin: Incobotulinum Toxin 100 units diluted in 1 ml of sterile 0.9% saline injected in the parotid (20 units, 0.2 ml each) and submandibular (30 units, 0.3ml each) glands of subjects
- Placebo: Sterile, preservative free 0.9% saline, 1 mL injected into the parotid (0.2 ml each) and submandibular (0.3ml each) glands .
Arm/Group | Incobotulinum Toxin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 2/9 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Incobotulinum Toxin (N=9) | Placebo (N=9)
chewing difficulty (Gastrointestinal disorders) | 1 (1) | 0 (0) — difficulty in chewing, a sensation of swelling inside the cheeks, a tendency to bite the inside of her cheeks and difficulty with motor control of the tongue, mild, resolved in 4-6 weeks without intervention
viscous saliva (Gastrointestinal disorders) | 1 (1) | 0 (0) — viscous, thick saliva, mild, resolved in 4-6 weeks without intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No